CLINICAL TRIAL: NCT07085858
Title: Study of the Preventive Effects and Mechanisms of Yeast β-Glucan on Upper Respiratory Tract Infections
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, lixiaoqin, Associate Professor, School of Public Health, Lanzhou University, LanZhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB25041502
Record Dates: First submitted 2025-07-04; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Upper Respiratory Tract Infections
Keywords: Upper respiratory tract infections; Yeast β-glucan
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yeast β-Glucan (Experimental): Participants in the intervention group will take yeast β-glucan capsules daily. Each capsule contains 250 mg of yeast β-glucan, along with an appropriate amount of maltodextrin and silicon dioxide. All participants in the intervention group will take two capsules once daily, swallowed with warm water after meals.
  Interventions: Dietary Supplement: yeast β-glucan
- placebo group (Placebo Comparator): Participants in the placebo group will take two placebo capsules once daily in the same manner. The placebo capsules are identical to the intervention capsules in form, taste, appearance, and packaging, but contain only maltodextrin and a small amount of silicon dioxide.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: yeast β-glucan — Participants in the intervention group will take yeast β-glucan capsules daily. Each capsule contains 250 mg of yeast β-glucan, along with an appropriate amount of maltodextrin and silicon dioxide. All participants in the intervention group will take two capsules once daily, swallowed with warm water after meals.
  Arms: Yeast β-Glucan
Dietary Supplement: placebo — Participants in the placebo group will take two placebo capsules once daily in the same manner. The placebo capsules are identical to the intervention capsules in form, taste, appearance, and packaging, but contain only maltodextrin and a small amount of silicon dioxide.
  Arms: placebo group

SUMMARY:
This study is designed as a randomized, double-blind, placebo-controlled human intervention trial targeting a population of university students with persistent allergic rhinitis (AR) symptoms. The primary objective is to evaluate the preventive effect and underlying mechanisms of yeast β-glucan on upper respiratory tract infections (URTIs), providing scientific evidence for the prophylactic use of prebiotics in high-risk populations.

All participants will be stratified by sex and body mass index (BMI), and then randomly assigned to either the yeast β-glucan group or the control group. During the 15-week study period-including a 1-week run-in phase, a 12-week intervention phase, and a 2-week follow-up phase-participants in the intervention group will take two yeast β-glucan capsules daily after meals, while the control group will take two placebo capsules with identical appearance, taste, and packaging.

Participants will be monitored daily for the occurrence of URTIs. In the event of an infection, the Wisconsin Upper Respiratory Symptom Survey (WURSS-24) will be used to assess symptom severity and duration. Medication use, including dosage, frequency, and timing, will also be recorded. Weekly follow-ups will assess changes in Total Nasal Symptom Score (TNSS), Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ), and adverse events. In addition, participants will undergo comprehensive follow-up assessments at Week 0 and Week 12, including TNSS and RQLQ questionnaires, a 3-day dietary intake survey, anthropometric measurements (e.g., height, weight, body fat percentage), and biological sample collection (blood, urine, and stool samples).

DETAILED DESCRIPTION:
Upper respiratory tract infections (URTIs) are acute mucosal infectious diseases caused by the invasion of respiratory mucosa by pathogens, which disrupt the mucosal barrier, activate the immune system, and trigger inflammatory responses. Clinical symptoms include nasal congestion, rhinorrhea, sore throat, cough, and hoarseness. Although URTIs are generally self-limiting, their high incidence, recurrence, and transmissibility-especially in crowded settings such as schools and workplaces-pose a significant public health burden. Allergic rhinitis (AR) is a chronic upper airway inflammatory disease mediated by immunoglobulin E (IgE), with typical symptoms such as nasal itching, sneezing, clear rhinorrhea, and nasal congestion. In AR patients, the nasal mucosa remains in a persistent inflammatory state, with impaired epithelial barrier function, reduced ciliary activity, and decreased local secretory IgA (sIgA) production. These alterations weaken the mucosal immune defense against viruses and bacteria, making AR patients more prone to recurrent URTIs. Furthermore, the seasonal onset of AR often coincides with peak URTI incidence, further compounding the risk of infection. Therefore, individuals with AR are considered a susceptible population for URTIs and are ideal targets for evaluating preventive interventions.

This study is designed as a randomized, double-blind, placebo-controlled human intervention trial among university students with persistent AR symptoms. The aim is to evaluate the preventive effect and underlying mechanisms of yeast β-glucan on URTIs, providing scientific evidence for the prophylactic application of prebiotics in high-risk populations. A total of 96 participants with persistent AR symptoms will be recruited and stratified by sex and BMI before being randomly assigned to either the yeast β-glucan group (n=48) or the placebo group (n=48). Blinding will be applied to both participants and investigators. Only the study designers will have access to the randomization codes. All intervention products and samples will be labeled with coded identifiers to prevent unblinding. If a participant experiences a serious adverse event related to the intervention, unblinding will be permitted, and the participant will be withdrawn from the study.

The yeast β-glucan used in this study is provided by Angel Yeast Co., Ltd. In 2010, China's Ministry of Health approved yeast β-glucan as a novel food ingredient for use in general food products, indicating its established safety. Nevertheless, adverse events will be closely monitored throughout the study and reported in accordance with ethical requirements.

During the intervention period, participants in the intervention group will take two yeast β-glucan capsules daily, each containing 250 mg of yeast β-glucan along with maltodextrin and silicon dioxide. The placebo group will receive identical capsules in terms of form, taste, appearance, and packaging, containing only maltodextrin and a small amount of silicon dioxide. All participants will take two capsules once daily after meals with warm water. Participants will be monitored daily for the occurrence of URTIs. If URTIs occur, the Wisconsin Upper Respiratory Symptom Survey (WURSS-24) will be used to assess symptom severity and duration, and medication use (number of doses, dosage, and timing) will be recorded. Weekly follow-ups will be conducted to assess Total Nasal Symptom Score (TNSS), Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ), and adverse events. At weeks 0 and 12, participants will complete questionnaire assessments (TNSS, RQLQ), a dietary intake survey, anthropometric measurements (e.g., height, weight, body fat percentage), and biological sample collection (blood, urine, and feces).

The primary outcome of this study is the incidence of URTIs. Secondary outcomes include: WURSS-24 (URTI symptom severity and duration), TNSS (nasal symptom score), RQLQ (quality of life assessment for rhinoconjunctivitis) ,Inflammatory cytokines (IFN-γ, IL-4, IL-10, IL-6, TNF-α) Serum biochemical markers(CRP, ALT/AST, BUN/Cr) and Fecal biomarkers (microbiota composition, SCFAs). Data will be analyzed using SAS 9.4 software. Continuous variables will be expressed as mean ± standard deviation; ordinal variables will be presented as percentages. Independent sample t-tests or Kruskal-Wallis tests will be used for continuous variables, and chi-square or Fisher's exact tests will be used for categorical variables. A p-value of < 0.05 will be considered statistically significant. For outcome variables with repeated measures at multiple time points (e.g., TNSS, inflammatory markers at weeks 0 and 12), a linear mixed-effects model (LMM) will be constructed to evaluate the effects of time, group, and their interaction, and to compare temporal trends between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 35 years;
2. Meeting the symptom criteria for persistent allergic rhinitis (AR) as defined in the Chinese Guidelines for Diagnosis and Treatment of Allergic Rhinitis (2022, Revised Edition): (1) Symptoms: Two or more of the following-paroxysmal sneezing, watery rhinorrhea, nasal itching, and nasal congestion-lasting continuously or cumulatively for at least 1 hour per day; ocular symptoms such as tearing, itching, and redness may also be present; (2) Persistent AR: Symptoms occur on ≥4 days per week and persist for ≥4 consecutive weeks;
3. No use of probiotics, prebiotics, synbiotics, antihistamines, corticosteroids, or immunosuppressants within 1 month prior to screening;
4. Willing and able to maintain usual physical activity levels and dietary patterns during the study;
5. Able and willing to sign the informed consent form voluntarily.

Exclusion Criteria:

1. Use of antibiotics, osmotic laxatives (e.g., magnesium sulfate, lactulose), anthraquinone-containing agents (e.g., rhubarb, aloe, senna), or gastrointestinal motility-promoting drugs (e.g., metoclopramide, domperidone, cisapride) within 1 month prior to screening;
2. Diagnosed with non-allergic rhinitis (e.g., vasomotor rhinitis, infectious rhinitis, hormonal rhinitis, drug-induced rhinitis), or with nasal polyps, severe nasal septum deviation, cerebrospinal fluid rhinorrhea, or aspirin-exacerbated respiratory disease (AERD);
3. Patients with uncontrolled allergic comorbidities, including sinusitis, otitis media, allergic asthma, or atopic dermatitis;
4. History of serious gastrointestinal diseases (e.g., severe diarrhea, inflammatory bowel disease), or gastrointestinal endoscopy within the past month;
5. Diagnosed with congenital genetic disorders, primary immunodeficiency diseases, severe systemic illnesses, or malignancies;
6. Influenza vaccination within the past 6 months;
7. Pregnant or lactating women, or women with plans to conceive during the study period.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Upper Respiratory Tract Infections (URTIs) | From enrollment to the end of intervention at 12 weeks

SECONDARY OUTCOMES:
Wisconsin Upper Respiratory Symptom Survey (WURSS-24) | From the onset of URTI symptoms up to 14 days after symptom onset. (through intervention completion, week 0 to week 12)
  The WURSS-24 is a 24-item validated questionnaire designed to assess the severity and duration of symptoms during upper respiratory tract infections (URTIs), as well as the impact on daily quality of life. Each item is rated on a 0-7 scale, with 0 indicating no symptoms or no impact, and 7 indicating the most severe symptoms or greatest impact. Higher total scores indicate worse outcomes. The total score ranges from 0 to 168.
Total Nasal Symptom Score (TNSS) | Each week through intervention completion (Week 0 to Week 12).
  A scoring system to evaluate the severity of four nasal symptoms: nasal itching, sneezing, rhinorrhea, and nasal congestion. Each symptom is rated on a scale of 0 to 3, with a total score ranging from 0 to 12. Higher scores indicate more severe symptoms.
Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | Each week through intervention completion (Week 0 to Week 12).
  A validated 28-item questionnaire covering seven domains: daily activities, sleep, nasal symptoms, ocular symptoms, emotional impact, practical problems, and environmental exposure. Each item is scored from 0 to 6; higher scores indicate greater impairment. Changes from baseline to post-intervention scores are used to evaluate improvements in quality of life.
IFN-γ | Baseline Week 12
  A signature cytokine of Th1-type immune responses, IFN-γ plays a critical role in activating macrophages, enhancing antigen presentation, and promoting cellular immunity. Fasting plasma levels of IFN-γ are measured using high-sensitivity ELISA kits.
IL-4 | Baseline Week 12
  IL-4 is central in the pathogenesis of allergic diseases such as asthma and allergic rhinitis, contributing to eosinophilic infiltration and IgE production. Fasting plasma levels of IL-4 are measured using high-sensitivity ELISA kits.
IL-10 | Baseline Week 12
  An anti-inflammatory cytokine that modulates immune responses by inhibiting the synthesis of pro-inflammatory cytokines. Fasting plasma levels of IL-10 are measured using high-sensitivity ELISA kits.
IL-6 | Baseline Week 12
  A pleiotropic cytokine involved in both pro-inflammatory and anti-inflammatory processes. It plays a role in acute-phase responses, B-cell differentiation, and chronic inflammation. Fasting plasma levels of IL-6 are measured using high-sensitivity ELISA kits.
TNF-α | Baseline Week 12
  TNF-α is a central pro-inflammatory cytokine involved in the initiation and amplification of inflammation. It plays a major role in systemic inflammation and is implicated in numerous inflammatory and autoimmune conditions. Fasting plasma levels of TNF-α are measured using high-sensitivity ELISA kits.
C-reactive protein (CRP） | Baseline Week 12
  CRP is an acute-phase reactant produced by the liver in response to inflammation. Elevated CRP levels serve as a sensitive, though non-specific, marker of systemic inflammatory activity. CRP levels are measured using an automated biochemical analyzer.
ALT/AST | Baseline Week 12
  ALT and AST are hepatic enzymes that reflect liver function. Elevated levels are indicative of hepatocellular injury or inflammation. ALT/AST levels are measured using an automated biochemical analyzer.
BUN/Cr | Baseline Week 12
  BUN and creatinine are metabolic waste markers used to evaluate kidney function. Abnormal levels may indicate renal impairment. The BUN/Cr ratio is useful in distinguishing between prerenal and renal causes of dysfunction. BUN/Cr levels are measured using an automated biochemical analyzer.
Gut Microbiota Composition | Baseline Week 12
  Fecal microbiota is analyzed using 16S rRNA gene amplicon sequencing to evaluate microbial diversity (α/β diversity), relative abundance of dominant taxa, and ecological shifts in response to intervention.
Short-chain fatty acids (SCFAs) concentration in feces | Baseline Week 12
  Measured by gas chromatography-mass spectrometry (GC-MS)
Fecal secretory immunoglobulin A (sIgA) levels | Baseline Week 12
  Measured by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health, Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT07085858/Prot_SAP_ICF_000.pdf